CLINICAL TRIAL: NCT02505178
Title: Examining the Feasibility and Effectiveness of Case Manager Delivered Problem Solving Therapy on Late Life Depression; an Open-label Prospective Pilot Study.
Brief Title: Examining the Feasibility and Effectiveness of Case Manager Delivered Problem Solving Therapy on Late Life Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Substantial changes were made to the study protocol and a new ethics application will be submitted.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other); Queen's University (Other)
Responsible Party: Principal Investigator, Akshya Vasudev, Akshya Vasudev MD, MRCPsych, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 106856
Record Dates: First submitted 2015-07-19; First posted 2015-07-22 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Depression
Keywords: Depression; Depressive Disorder; Depressive Disorder, Major; Mental Disorders; Mood Disorders; Behavioural Symptoms; Problem Solving Therapy
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major; Mental Disorders; Mood Disorders; Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Problem Solving Therapy (Experimental): Study participation will involve 9 study visits over a total of 12 weeks. This includes 5 sessions of Case Manager implemented PST over a period of 8 weeks (week 1, 3, 5, 7, and 9) and 4 assessment visits (baseline, week 4, week 8, and week 12).
  Interventions: Other: Problem Solving Therapy

INTERVENTIONS:
Other: Problem Solving Therapy — PST is a minimally invasive treatment. The five sessions of CM implemented PST will involve psychotherapy also known as talk therapy between the CM's and study participants in a group setting. Psychogeriatric interdisciplinary staff (CM's) i.e. psychiatric nurses, social workers who have been previously trained in PST will function in the roles of facilitator, cofacilitator and scribe. The roles can be shared amongst the professionals to build capacity in each role or maintained over time if so desired. Sessions will be approximately one-and-a-half to two hours in length and conducted at the Cherry Hill Mall library in London.

SUMMARY:
This study seeks to determine the feasibility and efficacy of a Problem Solving Therapy intervention for the treatment of late life depression (LLD). Participants diagnosed with LLD will participate in six sessions of Problem Solving Therapy, a form of talk-therapy, over a period of eight weeks. A Case Manager (CM) will lead the PST. The primary outcome measure is depression severity and will be measured throughout the study at weeks 0, 4, and 8. the secondary outcome measure is quality of life and will be measured at week 0 (pre-intervention) and week 12.

DETAILED DESCRIPTION:
In the elderly (i.e. individuals 60 years of age or older) major depressive disorder (MDD) is common occurring in 2-3% of the population and known as late life depression (LLD). LLD is both disabling and associated with a high mortality rate. Response to treatment of LLD using at least one antidepressant trial of adequate dose and duration is around 30-40%. Due to these suboptimal response rates, additional interventions should be tested and implemented to further alleviate the symptoms and severity of LLD.

It is common for individuals referred to geriatric psychiatry programs to live alone and have impaired independent mobility, which makes them more susceptible to depression as they are at a higher risk for social isolation. Best practice guidelines recommend using psychosocial therapies, which are effective in reducing symptoms of LLD, as the standard treatment for mild to moderate depression, either alone or in combination with medications. PST can be delivered to patients close to their homes making it ideal for treating seniors with limited mobility. The elderly are more likely to suffer from co-morbid conditions and be treated with multiple medications. Antidepressants are associated with serious adverse events, making psychosocial treatments especially important to the elderly who take more medications and are more likely to suffer comorbid conditions.

Problem-solving therapy (PST) is an established psychosocial therapy shown to be effective in treating depression and other mental disorders in adults of all ages. PST involves seven stages of problem resolution including a)identifying and clarifying the problem b)setting clear achievable goals c) brain-storming to generate solutions d) selecting a preferred solution and f) evaluation. Studies of PST in older adults have shown the treatment to be effective in reducing depression. PST has been successfully adapted to meet the needs of seniors with comorbid conditions and those with early dementia or cognitive impairment.

Despite the importance of psychotherapy interventions for older adults with MDD there is limited access to these treatments for seniors. At present, nurse case managers and social work case managers (CM) do not receive formal training in problem solving therapy. Since they often provide treatment for geriatric mental health outpatients, this limits access to treatments like PST. However, if CM's have formal training in PST, this treatment option can be made available to seniors that could benefit from such programs. To the best of the investigators' knowledge no study has evaluated the effects of CM trained to deliver PST for individuals with LLD in Canada, as such, this is the aim of the current investigation.

ELIGIBILITY:
Inclusion Criteria:

* Are of either gender and greater than 60 years of age.
* Reside in a community setting (either independent living environment or retirement home).
* Meet diagnostic criteria for major depressive disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V) criteria.
* Have a Hamilton Depression Rating Scale (HAMD) 17-item total score of >= 8 and < 24 at baseline.
* Have a Mini Mental Status Exam score of >= 20.
* Have adequate hearing and vision to be able to participate in Problem Solving Therapy.

Exclusion Criteria:

* Have suicidal ideation requiring inpatient admission to hospital for stabilization.
* Have an unstable medical condition requiring hospital admission.
* Have a life expectancy of less than 6 months or are currently receiving palliative care.
* Have psychotic symptoms.
* Have a lifetime history of bipolar disorder or schizophrenia.
* Are currently alcohol dependent or have another substance dependence.
* Are diagnosed with moderate to severe dementia.
* Are planning admission to a long-term care facility within next 6 months.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms | Baseline, week 4, and week 8
  Depression in study participants will be self rated on the Patient Health Questionnaire (PHQ-9)

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline and week 12
  Participants will complete a Short Form-12 to assess the change in their quality of life.
Change in Depression Symptoms- Clinician Rated | Baseline, Week 4 and Week 8
  Hamilton scale for Depression-17 item (HAM-D 17), as rated by a clinician trained to complete this scale
Change in Depression Symptoms- Overall improvement | Baseline, Week 4 and Week 8
  Clinical Global Impression- CGI, as rated by a clinician trained to complete this scale

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada